CLINICAL TRIAL: NCT00740077
Title: Bioavailability of Flavonoids and Phenolic Acids From Cranberry Juice Cocktail in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Jeffrey B. Blumberg, Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PV4266
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: cranberry; flavonoid; phenolic acid; phytochemical; bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Low calorie, sugar-free cranberry juice cocktail (54% juice) — Single-dose, 24 hour pharmacokinetic trial of 8 oz dose administered orally.

SUMMARY:
This is a single-dose, pharmacokinetic study investigating the bioavailability of flavonoids and phenolic acids from cranberry juice cocktail and their breakdown products (in vivo metabolites) in healthy, older adults. Our hypothesis is that the compounds will be poorly but rapidly absorbed from the intestines and found in plasma and urine in extensively metabolized forms. These compounds will be rapidly cleared from plasma. Substantial amounts of unabsorbed compounds will be found in the stools.

DETAILED DESCRIPTION:
Cranberries are a particularly rich source of phenolic acids and polyphenols, particularly flavonoids. Among the 20 most commonly consumed fruits in the American diet, cranberries have the highest total phenol content. Health benefits attributed to cranberries include the prevention of urinary tract infections and stomach ulcers as well as improved oral hygiene. These benefits appear to be due principally to the ability of cranberries to interfere with the adhesion of some bacteria to select cell types and surfaces.

Cranberries and cranberry constituents, including several phenolic and polyphenolic compounds, have also been shown to possess antibacterial, antiviral, anti-mutagenic, anti-carcinogenic, anti-tumorigenic, anti-angiogenic, and antioxidant activities. Most of this evidence is derived from in vitro studies and animal models. The limited number of human studies available indicate these phytochemicals are bioavailable and bioactive. However, more information is required on the bioavailability and metabolism of cranberry polyphenols, as well as on the relationship between cranberry dose and duration of use, to better understand their impact on risk factors for chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* BMI 18.5-29.9 kg/m2

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Use of any stomach acid-lowering medications
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 95 mm Hg
* Regular use of oral steroids
* Regular daily intake of 2 or more alcoholic drinks
* Illicit drug use
* No fish oil supplements (including cod liver oil) for one month prior to study admission
* No dietary supplements, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) or homeopathic remedies, for one month prior to study admission

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Levels of phenolic acids and flavonoids (including anthocyanins, flavanols, flavonols, and proanthocyanidins) and their in vivo metabolites in blood, urine, and feces following cranberry juice consumption. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Blumberg, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States